CLINICAL TRIAL: NCT02794753
Title: Cognitive Training in Patients With Trichotillomania (Hair-pulling Disorder)
Acronym: CTTTM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Stellenbosch (Other)
Collaborators: National Research Foundation, Singapore (Other Government); Medical Research Council, South Africa (Other); Stikland Psychiatric Hospital (Unknown)
Responsible Party: Principal Investigator, Derine Sandenbergh, Mrs Derine Sandenbergh, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UStellenbosch
Record Dates: First submitted 2016-05-27; First posted 2016-06-09 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Trichotillomania
Keywords: Trichotillomania; Hair-pulling Disorder; Cognitive Training; Neuroplasticity; Working Memory
MeSH Terms: conditions — Trichotillomania

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- True intervention (Experimental): Working memory training on computer 5 weeks 25 sessions (5 sessions per week) 50 minutes per session
  Interventions: Behavioral: Working memory training
- Active control (Active Comparator): Similar time spent playing on computer 5 weeks 25 sessions (5 sessions per week) 50 minutes per session
  Interventions: Behavioral: Game

INTERVENTIONS:
Behavioral: Working memory training
  Arms: True intervention
Behavioral: Game
  Arms: Active control

SUMMARY:
The principal aim of this study is to establish the impact of Cognitive Training in patients with primary Hair-pulling Disorder. Half of the participants will be training with the true training intervention and the other half with the active control intervention.

Study findings will also provide information on whether an internet based CT intervention, done at patients' homes, is feasible as a mode of treatment for HPD patients in SA.

DETAILED DESCRIPTION:
Introduction and conceptualization Hair-pulling disorder (HPD) has not received much attention in comparison to other psychiatric illnesses. Considering South African research, only a limited number of studies have focused on HPD with minimal focus on treatment interventions. Several treatments with regards to pharmacotherapy and psychotherapy have been developed and investigated. Evidence suggests limited efficacy of these treatments, thus there is a need for an intervention that shows better efficacy in symptom reduction with longer maintenance of treatment gains, whilst also being cost-effective and easily accessible. Studies have indicated that patients with HPD experience difficulty in working memory (WM), impulse control (IC) and emotion regulation (ER). The involvement of the frontoparietal circuitry, as well as frontal cortex, amygdalo-hippocampal formation and putamen have been specified in HPD. WM and ER circuitry are both based in the frontoparietal neural circuit, and thus training of WM shows potential to also address ER difficulties. An intervention focusing on WM training, may promise to address difficulties in IC and ER, and thus be appropriate in the treatment of patients with HPD. Cognitive training (CT) is a novel intervention that focuses on enhancing executive functioning and more specifically WM. WM tasks in CT also focus on the frontoparietal network which plays a role in ER, and therefore when this network is activated by executive functioning tasks, ER should improve. The positive impact of computerized cognitive training (CCT) on neuroplasticity in these indicated pathways have recently been acknowledged. Psychotherapeutic support might not be readily available or accessible to most people in developing countries, such as South Africa. Indeed, locally the physical distance from mental health centres and cost of individual sessions with health care professionals, are challenging - preventing patients finding the help that they need. CT can thus be a more accessible and cost-effective alternative. Cogmed Working Memory Training, an internet-based CT program, will be investigated for its efficacy in the treatment of HPD.

Purpose of the study: The principal aim of this project is to establish the impact of CT in patients with primary HPD. Study findings will also provide information on whether an internet based CT intervention, done at patients' homes, is feasible as a mode of treatment for HPD patients in SA. The proposed research will focus on the following objectives: To determine the effect of CT (25 sessions over 5 weeks) on WM, ER, IC and hair-pulling severity (HPS), in patients with HPD. To determine whether the effect of the true CT program on WM, ER, IC and HPS differed from that of the active control program. To determine whether effects are maintained at 3 months post-intervention. To qualitatively explore participants' subjective experience of the intervention process and responses to CT (in terms of WM, ER, IC and HPS).

It is hypothesised that after 5 weeks of CT, the treatment HPD group will show significant improvement in WM, ER, IC and significant reduction in HPS. The effect of the true CT program on WM, ER, IC and HPS will be significantly different from the active control group. During a 3-month follow-up evaluation, the HPD intervention group will have maintained reduction in symptoms after the treatment, compared to the active control HPD group. The treatment HPD group will generally be positive about the effects of CT on HPD and their functioning at post-intervention and 3-month follow-up and consider CT as easy to use and affordable.

Study design: The study design is a 5-week, 25-session intervention study with an active control, and 3-month follow-up evaluation. As a registered clinical psychologist, the principal investigator has the expertise to diagnose, do clinical interviews, and implement the psychometric battery pre and post intervention. Inclusion criteria is a primary diagnosis of HPD (DSM-5); Adults (18 years and older); Fluent in English; Access to the internet for the duration of their study participation. Exclusion criteria is any significant current DSM comorbidity; Montgomery-Asberg Depression Rating Scale (MADRS) Score > 20 to exclude patients with comorbid depressive syndromes; Previous exposure to cognitive training (previous 'brain training' games on cell phone and/or computer allowed). The criteria will be assessed during the screening procedure. Participants will enter the study as recruited and randomly assigned to the treatment or active control group. Participants entering the study will be randomized into the intervention or active control group, using a randomization list provided by the statistician. The intervention task (Cogmed QM) and the placebo (Jigsaw Puzzles) differ significantly. The principal investigator will not be blind to the group that the participants are in, whereas the participants will be blind to their group inclusion. It is aimed to achieve a sample size of at least 40 (20 treatment, 20 active control). This is comparable to group sizes in other HPD treatment studies. The research method is based in embedded theory design, utilizing both quantitative and qualitative components. The benefit of this hybrid approach is to be able to investigate and describe subject matter with statistical power, as well as being able to comment on the participant's experience, thus creating a richer and more holistic description of the research theme. The quantitative research consists of the pre- and post intervention assessment battery, 3-month follow-up evaluation and continuous information provided by the treatment intervention (Cogmed). The qualitative data analysis will be done on semi-structured interviews, as part of the pre- and post assessment battery and 3-month follow-up evaluation. Pre- and post intervention data collection will be done by the principal investigator by means of the assessment battery including both quantitative and qualitative measures. Statistical analysis will be conducted using mixed model repeated measures ANOVA, which is most suitable for dealing with possible lost to follow-up. Patients in the study will be treated as random effects (randomly selected from a larger population). Treatment (intervention vs placebo) and time (pre, post, 3 months) will be treated as fixed effects. The treatment*time interaction effect will be the primary effect of investigation because it tests whether the change over time is the same for the two groups. If the intervention has a different effect to the placebo, then this interaction effect should be significant. Post hoc testing will be done using Fisher Least Significant Difference (LSD) testing. Normality assumptions will be checked for all analyses and appropriately dealt with if necessary, based on the nature of the data. A 5% significance level will be used as guideline for significant results. The qualitative data will be analysed using an interpretative phenomenological approach (TerreBlanche, Durrheim, & Kelly, 2010), utilizing a qualitative data analysis software program, Atlas.ti.

Anticipated benefits and risks: CT has not been investigated as a treatment intervention for HPD and reduction of HPS cannot be guaranteed. However, HPS may reduce during the true CT program. Participants, who are part of the placebo group, will get the opportunity to access the true CT program on completion of the study. Except for the fact that they might not be in the treatment group for the duration of the study due to randomization, there are no known risks involved in participation.

Ethical Considerations: The study procedures, risks and benefits will be communicated in lay terminology to all participants (verbally and in writing) in Afrikaans or English. All data collected will be kept strictly confidential and study results made public and published without compromising confidentiality. The demographics questionnaire will be removed from the questionnaire pack to ensure that the completed questionnaires and the demographic details cannot be linked. Personal identifying details such as the name and contact information will not be recorded on the electronic database. All participants will be allocated a unique study code on the electronic database. Identifiers linked to a study code will be kept in a separate, password protected file. Only the principal investigator will have access to this information. It will be clearly indicated that the participant is free to withdraw participation from this trial, without consequence. Participating individuals will incur no costs.

ELIGIBILITY:
Inclusion Criteria:

* 18 year or older
* Diagnosis of HPD
* Proficient in English
* MADRS score < 20

Exclusion Criteria:

* Younger than 18 years.
* Doesn't have HPD.
* Has a serious medical condition or a previous head injury (this may impact on findings).
* Diagnosis of depression, obsessive-compulsive disorder, substance use disorder or any other significant mental disorder (other than HPD).
* Cannot understand or speak English (many of the tests used in the project, as well as the chosen intervention, is only available in English).
* Have received cognitive training before (previous 'brain training' games on cell phone and/or computer allowed).
* Do not have access to a laptop or desktop computer with reliable internet connection at home.
* On a psychotropic medication for less than 6 weeks before starting the trial. However, will remain eligible if receiving treatment at time of screening, provided the following restrictions are met: You are only receiving a single psychotropic medication & the medication being treated with, have been taken at a steady dose, for at least 8 weeks and effect stabilizing according to psychiatrist.
* You are not undergoing therapy. However you will remain eligible if you are receiving treatment from a psychologist or other mental health clinician at time of screening and continue to do so for the duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Hair-pulling symptoms from baseline to immediately after 5 weeks of cognitive training / placebo, measured using the Massachusetts General Hospital - Hair-pulling Scale (MGH-HPS). | Pre-intervention (prior to starting the training / placebo) to post-intervention (immediately after the 5 weeks training).
Change in Hair-pulling symptoms from immediately after 5 weeks of cognitive training / placebo to 3 months after completion of cognitive training / placebo, measured using the Massachusetts General Hospital - Hair-pulling Scale (MGH-HPS). | Post-intervention (immediately after the 5 weeks training) to 3 months Post-intervention (3 months after the training / placebo has been completed)

SECONDARY OUTCOMES:
Change in Emotional regulation from baseline to immediately after 5 weeks of cognitive training / placebo, measured using the Affective Regulation Scale (ARS) and the Difficulty in Emotional Regulation Scale (DERS). | Pre-intervention (prior to starting the training / placebo) to post-intervention (immediately after the 5 weeks training).
Change in Emotional regulation from immediately after 5 weeks of cognitive training / placebo to 3 months after completion thereof, measured using the Affective Regulation Scale (ARS) and the Difficulty in Emotional Regulation Scale (DERS) | Post-intervention (immediately after the 5 weeks training) to 3 months Post-intervention (3 months after the training / placebo has been completed).
Change in ability for Impulse control baseline to immediately after 5 weeks of cognitive training / placebo, measured using the Barratt Impulsiveness Scale (BIS-11) and Stroop Color and Word Test - Adult Version (SCWT-A). | Pre-intervention (prior to starting the training / placebo) to post-intervention (immediately after the 5 weeks training).
Change in ability for Impulse control from immediately after 5 weeks of cognitive training / placebo to 3 months after completion thereof, measured using the Barratt Impulsiveness Scale (BIS-11) and Stroop Color and Word Test - Adult Version (SCWT-A) | Post-intervention (immediately after the 5 weeks training) to 3 months Post-intervention (3 months after the training / placebo has been completed
Change in Working memory, from baseline to immediately after 5 weeks of cognitive training / placebo, measured by Letter Number Sequencing (LNS) and Digit Span (DS) - both subtests from the Wechsler Adult Intelligence Scale 3rd edition (WAIS-III). | Pre-intervention (prior to starting the training / placebo) to post-intervention (immediately after the 5 weeks training).
Change in Working memory from immediately after 5 weeks of cognitive training / placebo to 3 months after completion thereof, measured using the Letter Number Sequencing (LNS) and Digit Span (DS) - subtests from the WAIS-III. | Post-intervention (immediately after the 5 weeks training) to 3 months Post-intervention (3 months after the training / placebo has been completed).

CONTACTS AND LOCATIONS:
Overall Officials: Derine Sandenbergh, MSc, Principal Investigator — Senior clinical psychologist / Lecturer
Locations (1):
- Stellenbosch University, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Findings will be made available in dissertation, as well as published in articles.